CLINICAL TRIAL: NCT03218462
Title: Effect of Sensory Adapted Dental Environment on Dental Anxiety of Children With Intellectual and Developmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20009272
Record Dates: First submitted 2017-06-27; First posted 2017-07-14 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Developmental Disability; Intellectual Disability; Dental Anxiety
Keywords: sensory adapted environment; pediatric dentistry; oral health; Developmental Disability; Intellectual Disability; dental anxiety; autism spectrum
MeSH Terms: conditions — Developmental Disabilities; Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Sensory adapted dental environment (SADE) at first exam (visit 1)
  Interventions: Behavioral: Sensory Adapted Dental Environment (SADE)
- Group 2 (Experimental): Sensory adapted dental environment (SADE) at recall exam (visit 2)
  Interventions: Behavioral: Sensory Adapted Dental Environment (SADE)

INTERVENTIONS:
Behavioral: Sensory Adapted Dental Environment (SADE) — No fluorescent room lights, solar projector on ceiling, regular dental x-ray apron laying on patient, quiet music playing in background

SUMMARY:
Children with intellectual/developmental disabilities (ID/DD) will experience less dental anxiety and cooperate better in a Sensory Adapted Dental Environment (modified visual, sensory, and somatosensory stimuli in a regular dental setting) than in a regular dental environment (RDE).

DETAILED DESCRIPTION:
The aim of this pilot study is to determine the effect of sensory adapted dental environment (SADE) on reducing dental anxiety of children with intellectual and/or developmental disabilities (ID/DD). With the growing number of children diagnosed with ID/DD and their inclusion in the community, there are more opportunities for dentists to encounter this population for their routine oral health care. If improvement in dental anxiety and behavior is evident from the study, as other pilot studies have suggested, it can be applied as one of clinical tools for treating children with ID/DDs. Furthermore, utilization of a SADE in clinical training of pediatric dentists or general dentists can improve clinicians' comfort level in managing behavior of individuals with ID/DD. This will encourage more clinicians to provide care and address the unmet oral health needs of this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Children with intellectual and/or developmental disabilities

Exclusion Criteria:

* No specific diagnosis
* Parents/guardians have limited English proficiency

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Behavior during initial dental exam | Day 1
  Measured using Frankl Scale for pediatric dentistry, with 1=definitely negative and 5=definitely positive
Behavior during recall exam | 3 months
  Measured using Frankl Scale for pediatric dentistry, with 1=definitely negative and 5= definitely positive

SECONDARY OUTCOMES:
Physiologic outcomes (oxygen saturation) during initial exam | Day 1
  Measured every 5 minutes during the exam (up to one hour)
Physiologic outcomes (oxygen saturation) during recall exam | 3 months
  Measured every 5 minutes during the exam (up to one hour)
Physiologic outcomes (hearts rate) during initial exam | Day 1
  Measured every 5 minutes during the exam (up to one hour)
Physiologic outcomes (hearts rate) during initial exam | 3 months
  Measured every 5 minutes during the exam (up to one hour)
Patient cooperation during initial exam | Day 1
  Assessed by parent/caregiver with post treatment written survey
Patient cooperation during recall exam | 3 months
  Assessed by parent/caregiver with post treatment written survey

CONTACTS AND LOCATIONS:
Overall Officials: Patrice B Wunsch, DDS, MS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No